CLINICAL TRIAL: NCT06863246
Title: Influence of Cognitive Load on Postural Control in People With Chronic Obstructive Pulmonary Disease
Brief Title: Postural Control in Chronic Obstructive Pulmonary Disease
Acronym: NEUROTIGUE P
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Université de Toulon (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-006
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Postural control; Variability; Non-linear; Cognitive task; Static balance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COPD: Patients with chronic obstructive pulmonary disease
  Interventions: Other: Evaluation of cognitive task on static balance; Other: Evaluation of visual feedback on static balance
- Control participants: Healthy individuals
  Interventions: Other: Evaluation of cognitive task on static balance; Other: Evaluation of visual feedback on static balance

INTERVENTIONS:
Other: Evaluation of cognitive task on static balance — Static balance with and without cognitive task (i.e., 1-back task)
Other: Evaluation of visual feedback on static balance — Static balance with and without visual feedback (i.e., eyes closed and open).

SUMMARY:
Postural control impairment is common in people with COPD (pwCOPD), which can increase the risk of falls and affect quality of life. However, the majority of existing studies examine this postural control in isolation, without taking into account the cognitive demands that occur during activities of daily living during which individuals are often required to perform a mental task while maintaining their balance. This research aims to fill this gap by studying how a cognitive task can influence postural control in pwCOPD. We hypothesized an impaired postural control in pwCOPD compared to healthy individuals, which would be exacerbated in presence of a cognitive task.

DETAILED DESCRIPTION:
This observational study is based on the analyses of data (center of pressure displacement) recorded during the first visit of NEUROTIGUE study (NCT04028973).

Center of pressure (COP) displacement were recorded during 60s of static balance in four conditions (random order) :

* Eyes open without cognitive task
* Eyes open with cognitive task
* Eyes closed without cognitive task
* Eyes closed with cognitive task The cognitive task used was a working memory task : the 1-back task. COP displacement will be assess using a conjunction of parameters to provide a comprehensive understanding of postural control (e.g., amplitude, standard deviation, non-linear approaches).

ELIGIBILITY:
Inclusion Criteria:

COPD patients :

* GOLD II - III or IV
* FEV1 <80% of predicted values
* Men and women aged 40 years and over
* French-speaking participant
* BMI <30 kg / m²
* Stable condition (i.e. without exacerbation) for more than 15 days
* Able to express their consent in writing prior to any participation in the study
* Affiliates or beneficiaries of a social security
* Minimum score of 26 on the MMSE questionnaire of 3 months or less

Healthy volunteers :

* Men and women aged 40 years and over
* French-speaking participant
* BMI <30 kg / m²
* No known chronic respiratory, cardiovascular, metabolic, renal or neuromuscular pathologies
* Able to express their consent in writing prior to any participation in the study
* Affiliates or beneficiaries of a social security
* Minimum score of 26 on the MMSE questionnaire of 3 months or less

For all participants :

-Subject who has not objected to the reuse of data collected

Exclusion Criteria:

* COPD patients :
* Alcoholism, i.e. > 21 glasses a week for men and >14 glasses a week for women
* Psychiatric pathologies or antecedent of behavioral disorders
* Patients treated with oral or systemic corticosteroids (> 0.5 mg / kg / day for > 7 days)
* Contraindication to the application of a magnetic field (i.e. right hip arthroplasty, pelvic / abdominal surgeries)
* Severe vision or hearing problems not corrected
* Patient oxygen dependent
* Patients in exclusion period from another research protocol
* Pregnant women (known pregnancy) or lactating women
* Patient deprived of liberty by a judicial or administrative decision
* Patient subject to a legal protection measure or unable to express their consent
* Patient who is not sufficiently fluent in reading and understanding the French language to be able to consent to participate in the study
* Patient unable to follow study procedures and to respect visits throughout the study period
* Person with a medical history that, in the opinion of the investigator, could interfere with the results of the study
* Any condition that, in the opinion of the investigator, could increase and compromise the safety of the person in the event that he / she participates in the study
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the aims of the study

Healthy volunteers:

* Alcoholism, i.e. > 21 glasses a week for men and >14 glasses a week for women
* Psychiatric pathologies or antecedent of behavioral disorders
* Patients treated with oral or systemic corticosteroids (> 0.5 mg / kg / day for > 7 days)
* Contraindication to the application of a magnetic field (i.e. right hip arthroplasty, pelvic / abdominal surgeries)
* Severe vision or hearing problems not corrected
* Subjects in exclusion period from another research protocol
* Pregnant women (known pregnancy) or lactating women
* Regular physical activity with a frequency greater than 3 sessions per week
* Participant deprived of liberty by a judicial or administrative decision
* Participant subject to a legal protection measure or unable to express their consent
* Participant who is not sufficiently fluent in reading and understanding the French language to be able to consent to participate in the study
* Participant unable to follow study procedures and to respect visits throughout the study period
* Person with a medical history that, in the opinion of the investigator, could interfere with the results of the study
* Any condition that, in the opinion of the investigator, could increase and compromise the safety of the person in the event that he / she participates in the study
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the aims of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in NEUROTIGUE study (NCT04028973)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Difference of the range of COP displacement between groups and experimental conditions | 10 minutes
  Range of COP displacement correspond to the maximal amplitude of the path of COP in anteroposterior and mediolateral directions.

SECONDARY OUTCOMES:
Difference of Sample Entropy (SampEn) of COP displacement between groups and experimental conditions | 10 minutes
  SampEn is a non-linear approach allowing to quantify the regularity of COP displacement in anteroposterior and mediolateral directions.
Difference of total COP displacement between groups and experimental conditions | 10 minutes
  The total COP displacement corresponds to the total distance covered by the COP during a recording period.
Difference of area of COP displacement between groups and experimental conditions | 10 minutes
  Area of COP displacement represents the area covered by COP during a recording period.

OTHER OUTCOMES:
Difference of mean COP position between groups and experimental conditions | 10 minutes
  Difference of mean COP position between groups and experimental conditions
Difference of the mean speed of COP displacement between groups and experimental conditions | 10 minutes
  Difference of the mean speed of COP displacement between groups and experimental conditions

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Vallier, MD, PHD, Study Director — Université de Toulon
Locations (1):
- Université de Toulon - Laboratoire J-AP2S, Toulon, VAR, France

IPD SHARING:
Plan to Share IPD: Undecided